CLINICAL TRIAL: NCT01296867
Title: Corneal Asphericity Adjustment (Q Adjustment) in Myopic and Hyperopic Patients Undergoing Refractive Correction With Excimer Laser
Status: Completed | Type: Observational
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Eleftherios Paschalis / PhD, Eye Institute of Thrace / Democritus University
Other Study IDs: Q-value
Record Dates: First submitted 2011-02-15; First posted 2011-02-16 (Estimated); Last update posted 2011-02-16 (Estimated); Status verified 2011-02

CONDITIONS: Myopia; Hyperopia
Keywords: Laser ablation algorithms; Excimer laser; Refractive correction; Corneal Asphericity Adjustment
MeSH Terms: conditions — Myopia; Hyperopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To study the postoperative results in myopic and hyperopic eyes treated with two different laser ablation algorithms (STD and F-CAT), both FDA approved.

ELIGIBILITY:
Inclusion Criteria:

* Myopic and hyperopic eyes eligible for LASIK or PRK refractive correction
* Central corneal thickness more than 500 micrometers

Exclusion Criteria:

* Topographies of less than 55% of successful total sampled area and eyes exhibiting asphericity variations, in either the horizontal or the vertical axis, greater than 0.2
* Corneal scarring
* Cataract surgery
* Corneal ulceration
* Topographical abnormalities

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Forty eight myopic (24 patients) and 24 hyperopic eyes (12 patients)
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2006-03; Primary Completion 2009-03 (Actual); Study Completion 2009-05 (Actual)